CLINICAL TRIAL: NCT06402201
Title: Phase 1, First-in-Human Study to Assess the Safety, Tolerability and Anti-tumor Activity of CDR404 in HLA-A*02:01 Participants With MAGE-A4 Expressing Solid Tumors
Brief Title: First in Human Study of CDR404 in HLA-A*02:01 Participants With MAGE-A4 Expressing Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CDR-Life AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDR404-001
Record Dates: First submitted 2024-04-25; First posted 2024-05-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Select Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: IV dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CDR404 (Experimental): Dose escalation
  Interventions: Biological: CDR404

INTERVENTIONS:
Biological: CDR404 — IV infusions

SUMMARY:
CDR404 is a highly potent and specific T-cell engaging bispecific and bivalent antibody designed for the treatment of cancers positive for the tumor-associated antigen melanoma-associated antigen 4 (MAGE-A4). This is a first-in-human study designed to evaluate the safety, tolerability, and preliminary anti-tumor activity of CDR404 in adult patients who have the appropriate germline human leukocyte antigen HLA-A*02:01 tissue marker and whose cancer is positive for MAGE-A4.

DETAILED DESCRIPTION:
The CDR404-001 Phase 1 study will enrol patients with locally advanced, unresectable or metastatic tumors expressing MAGE-A4, which include advanced solid tumors, and will be conducted in multiple phases:

1. To identify the maximum tolerated dose (MTD) and pharmacologically effective dose range (PEDR) for CDR404
2. To assess preliminary evidence of anti-tumor activity of CDR404
3. To characterise the pharmacokinetics of CDR404
4. To characterise the immunogenicity of CDR404
5. To assess translational biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. HLA-A*02:01 positive
3. MAGE-A4 positive tumor
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) [ECOG PS] 0 or 1
5. Selected advanced solid tumors
6. Relapsed from, refractory to, or intolerant of standard therapy
7. Measurable disease per RECIST v1.1
8. Adequate organ function
9. If applicable, must agree to use highly effective contraception

Exclusion Criteria:

1. Symptomatic or untreated central nervous system metastasis
2. Inadequate washout from prior anticancer therapy
3. Significant ongoing toxicity from prior anticancer treatment
4. Recent surgery
5. Clinically significant cardiac disease
6. Active infection requiring systemic antibiotic treatment
7. Human immunodeficiency virus (HIV) at risk of acquired immunodeficiency syndrome (AIDS)-related outcomes
8. Active hepatitis B virus (HBV) or hepatitis C virus (HBC)
9. Ongoing treatment with systemic steroids or other immunosuppressive therapies
10. Significant secondary malignancy
11. History of chronic or recurrent active autoimmune disease requiring treatment
12. Uncontrolled intercurrent illness
13. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of dose limiting toxicities (DLTs) | From first dose to DLT period (21 days)
  per Protocol
Incidence and severity of (serious) adverse events ([S]AEs) | From first dose to 90 days after the last dose
  AEs, SAEs
Anti-tumor response: Overall Response Rate (ORR) | From first dose until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  per RECIST 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | From first dose until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  per RECIST 1.1
Duration of response (DOR) | From first dose until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  per RECIST 1.1
Progression-free Survival (PFS) | From first dose until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  per RECIST 1.1
Overall Survival (OS) | From first dose until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  per RECIST 1.1
Maximum serum concentration of CDR404 (Cmax) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Time to maximum serum concentration of CDR404 (Tmax) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Trough serum concentration of CDR404 (Ctrough) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Half-life of CDR404 (t1/2) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Area under the CDR404 serum concentration over time curve (AUC0-T) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  to the end of the dosing interval following single and multiple dose administration
Volume of CDR404 distribution (Vd) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Average serum concentration of CDR404 (Cavg) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Serum drug levels of CDR404 at steady state (CL) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Accumulation ratio of CDR404 (Rac) | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
  following single and multiple dose administration
Immunogenicity | From first dose until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Incidence of detectable anti-CDR404 antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (4):
  - University of Miami, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Providence Cancer Institute, Portland, Oregon
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, UCL Ouvain, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Rigshospitalet, Copenhagen, Denmark
- Italy (2):
  - Istituto Clinico Humanitas, Milan
  - Isituto Europeo di Oncologia (IEO), Milan
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat (ICO), Barcelona
  - Hospital 12 de Octubre, Madrid
  - START Madrid, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Instituto de Investigacion Sanitaria (INCLIVA), Valencia

IPD SHARING:
Plan to Share IPD: No